CLINICAL TRIAL: NCT01534325
Title: Efficacy Study of SD Device for Overweight and Obesity Treatment
Brief Title: Efficacy Study for SD Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beck Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BeckMedical-001
Record Dates: First submitted 2012-01-12; First posted 2012-02-16 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Study arm (Experimental): The Arm who uses the real study device Daily use of SD device
  Interventions: Device: SD
- Control Arm (Sham Comparator): Daily use of Sham comperator
  Interventions: Device: Control
- Staudy2 arm (Experimental): Uses the under study device in a different time frames Daily use of SD device in a different time frames than of Study Arm
  Interventions: Device: SD

INTERVENTIONS:
Device: SD — The participants in the study receive basic nutrition guidance by MD and clinical dietician and make daily use of the device under study (called SD). During the 13 weeks study period, the participants get to meet clinical dietician/MD once in every 2 weeks for guidance and supervision and for on -going monitoring of physical parameters such as body weight and waist circumference.
  The use of the SD device is done by study participants during the day every day throughout the study period. The device under study can be easily used by the participants themselves in their regular environment and does not require professional assistance.
  The device under study is expected to affects the satiety, energy homeostasis and metabolic control centers in the brain and by that to reduce food intake and lead to weight loss.
  The device under study is a device- not a medication and not a surgical procedure, and it does not involve any of such elements.
  Arms: Study arm
Device: Control — The participants in the Control arm of the study receive basic nutrition guidance by MD and clinical dietician and make daily use of the placebo. During the 13 weeks study period, the participants get to meet clinical dietician/MD once in every 2 weeks for guidance and supervision and for on -going monitoring of physical parameters such as body weight and waist circumference.
  The use of the placebo is done by the control study participants during the day every day throughout the study period. The placebo can be easily used by the participants themselves in their regular environment and does not require professional assistance.
  Arms: Control Arm
Device: SD — The participants in the study receive basic nutrition guidance by MD and clinical dietician and make daily use of the device under study (called SD). During the 13 weeks study period, the participants get to meet clinical dietician/MD once in every 2 weeks for guidance and supervision and for on -going monitoring of physical parameters such as body weight and waist circumference.
  The use of the SD device is done by study participants during the day every day throughout the study period. The device under study can be easily used by the participants themselves in their regular environment and does not require professional assistance.
  The device under study is expected to affects the satiety, energy homeostasis and metabolic control centers in the brain and by that to reduce food intake and lead to weight loss.
  The device under study is a device- not a medication and not a surgical procedure, and it does not involve any of such elements.
  Arms: Staudy2 arm

SUMMARY:
The purpose of this study is to determine whether the SD unique device is effective in treatment of overweight and obesity.

DETAILED DESCRIPTION:
Obesity and Overweight had become the number 1 health concern of the modern world. Over 1 Billion people worldwide are overweight or obese. Those who suffer from overweight or obesity are exposed to other severe illnesses such as: diabetes, cardiovascular disease and cancer.

Only few drugs and surgeries are currently available as approved treatments for those who wish to reduce weight.

The purpose of this study is to determine whether the SD unique medical device, is effective in treatment of overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30-41.99
* AGE 18-65 years

Exclusion Criteria:

* Pregnant Women,
* Type I and II diabetes,
* People with disfunctioning of thyroid gland
* Hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-07; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Body Weight | once in every two weeks up to 13 weeks for each participant
  Each participant's body weight will be measured at his/her beginning of the trial. This measure will become the participant's body weight base-line. Once in every 2 weeks the body weight will be taken again and will be compared to base-line and to previous body weight measures of the participant taken during the study.

SECONDARY OUTCOMES:
Change from Baseline in Waist Circumference | once in every two weeks up to 13 weeks for each participant
  Each participant's Waist circumference will be measured at his/her beginning of the trial. This measure will become the participant's Waist circumference base-line. Once in every 2 weeks the Waist circumference will be taken again and will be compared to base-line and to previous Waist circumference measures of the participant taken during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Dror Dicker, MD, Principal Investigator — Rabin Medical Center
Locations (2):
- Israel (2):
  - Emek Medical Center, Afula
  - Rabin Medical Center, Petah Tikva